CLINICAL TRIAL: NCT06415799
Title: Verification of Investigational Pulse Oximetry Devices With the Abbreviated Sensor Line in Adult Volunteers
Brief Title: OM2 Abbreviated Sensor Verification
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT23027OM2VAB
Record Dates: First submitted 2024-04-19; First posted 2024-05-16 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-04

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Healthy Volunteers

SUMMARY:
The verification of an investigational pulse oximetry board to verify pulse rate and saturation accuracy over a specified saturation range in diverse populations.

DETAILED DESCRIPTION:
To verify the SpO2 and pulse rate accuracy in comparison to reference-standard blood measurements. To achieve paired observations of SpO2 and SaO2 values over the specified SpO2 accuracy range of the prototype pulse oximeter on a group of healthy adult volunteers. The fraction of inspired oxygen (FiO2) delivered to test subjects is varied to achieve a series of targeted steady-state saturation periods. In this study, the investigational pulse oximetry PCBA system saturation measurements will be compared to saturation measurements made by a multi-wavelength CO-oximeter, taken from arterial blood samples from a diverse pool of healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 50 years of age
2. Subject is willing and able to comply with study procedures and duration
3. Subject is willing to sign an informed consent
4. Subject weighs >40kg
5. Subject is a non-smoker or has not smoked within 2 days prior to the study
6. Cleared same day health assessment form and health screening
7. Successful perfusion index ulnar/ulnar+radial ratio test showing adequate collateral blood flow.

Exclusion Criteria:

1. Subject is considered as being morbidly obese (defined as BMI >39.5)
2. Compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the sites utilized)
3. Females of childbearing potential who are pregnant, who are trying to get pregnant, or who have a urine test positive for pregnancy on the day of the study
4. Subjects with COHb levels >3% as assessed by CO-Oximetry during the procedure
5. tHb < 10 g/dl as assessed by CO-Oximetry during the procedure
6. MetHb ≥ 2% as assessed by CO-Oximetry during the procedure
7. Subjects with known respiratory conditions such as:

   1. uncontrolled / severe asthma
   2. flu or influenza type infection
   3. pneumonia / bronchitis
   4. shortness of breath / respiratory distress
   5. unresolved respiratory or lung surgery
   6. emphysema, COPD, lung disease
   7. recent COVID (last 2 months)
8. Subjects with known heart or cardiovascular conditions such as:

   1. hypertension: systolic >140mmHg, or Diastolic >90mmHg on 3 consecutive readings
   2. have had cardiovascular surgery
   3. chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
   5. previous heart attack
   6. blocked artery
   7. unexplained shortness of breath
   8. congestive heart failure (CHF)
   9. history of stroke
   10. transient ischemic attack
   11. carotid artery disease
   12. myocardial ischemia
   13. myocardial infarction
   14. cardiomyopathy
   15. implantable active medical device such as pacemaker or automatic defibrillator
9. Self-reported health conditions as identified in the Health Assessment Form

   1. diabetes
   2. uncontrolled thyroid disease
   3. kidney disease / chronic renal impairment
   4. history of seizures (except childhood febrile seizures)
   5. epilepsy
   6. history of unexplained syncope
   7. recent history of frequent migraine headaches
   8. recent symptomatic head injury, within the last 2 months
   9. cancer requiring chemotherapy, radiation, or current treatment
   10. subjects with known clotting disorders
   11. history of bleeding disorders or personal history of prolonged bleeding from injury
   12. history of blood clots
   13. hemophilia
   14. sickle cell trait or disease
   15. current use of blood thinner: prescription or daily use of aspirin
   16. subjects with Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
   17. participants with severe allergy to iodine (only applicable if iodine is used)
   18. subjects with prior or known severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain) or heparin
   19. arterial cannulation within the last 30 days prior to study date, (this may exclude only one radial artery site, left or right)
   20. history of clinically significant complications from previous arterial cannulation
   21. unwillingness or inability to remove colored nail polish or colored artificial nails other than clear from test digits
   22. other known health condition, upon disclosure in Health Assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Male or Female volunteers age 18 to 50 years, weighing greater than 40kgs. Volunteers must be non-smokers or not smoked within 2 days prior to the study. Cleared a same day health assessment form and health screen to ensure none of the exclusion criteria was met. With a successful perfusion index ulnar/ulnar+radial ratio test showing adequate collateral blood flow.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Verification of Saturation Accuracy | 2.5 hours
  Saturation accuracy in a diverse subject population over a specified saturation range.
  The acceptance criteria for the investigational Pulse Oximetry PCBA system, SpO2 across the saturation range of 70-100%:
  SpO2 Max-A ±2% (ARMS) OxySoft-N ±2% (ARMS) Max-Fast ±2% (ARMS) FlexMax ±2.5%(ARMS) DS-100A ±3% (ARMS) D-YS ±3% (ARMS)
Verification of Pulse Rate | 2.5 hours
  Pulse rate in a diverse subject population over a specified saturation range.
  The acceptance criteria for pulse rate from 20-250 BPM over a specified saturation range of 70-100%:
  Pulse Rate Max-A ≤3% BPM (ARMS) OxySoft-N ≤3% BPM (ARMS) Max-Fast ≤3% BPM (ARMS) FlexMax ≤3% BPM (ARMS) DS-100A ≤3% BPM (ARMS) D-YS ≤3% BPM (ARMS)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, Principal Investigator — Element Labs
Locations (1):
- Element, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No